CLINICAL TRIAL: NCT02004080
Title: CREACTIVE - Collaborative REsearch on ACute Traumatic Brain Injury in intensiVe Care Medicine in Europe
Acronym: CREACTIVE
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Collaborators: European Commission (Other); Semmelweis University (Other); Medical University of Warsaw (Other); General Hospital of Novo mesto (Other); Univerzitetni Klinikni Center Ljubljana (Unknown); University of Nicosia (Other); Ben-Gurion University of the Negev (Other); University of Crete Medical School - University Hospital of Heraklion (Unknown); Orobix Srl (Unknown)
Responsible Party: Sponsor
Other Study IDs: 602714
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Brain Injuries, Traumatic
Keywords: TBI; ICU; Comparative Effectiveness Research
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood samples day 1 and 5 from ICU admission.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TBI admitted to ICU: Intensive Care treatment
  Interventions: Other: Intensive Care treatment

INTERVENTIONS:
Other: Intensive Care treatment — intensive care treatment

SUMMARY:
CREACTIVE is a large-scale observational cohort study concerning Traumatic Brain Injury (TBI) care in the ICU setting

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is among the leading causes of death and disability and the main cause of death among the under-45s. Most patients with moderate to severe TBI are admitted to intensive care units (ICUs).

The 'PROmoting patient SAFEty and quality improvement in critical care' ICU network was recently established in 6 European countries through European Union funding (PHEA 2007331), and has continued to collect high-quality data beyond the grant duration. In 2012, 242 ICUs had joined 'PROmoting patient SAFEty and quality improvement in critical care', recruiting a total of 85,965 patients. Of these ICUs, 180 admitted at least one TBI patient, totaling more than 3,300 cases. Hence, the network is expected to enroll 7-9,000 moderate-to-severe TBI patients in 4 years, in about 125 participating ICUs. The 'PROmoting patient SAFEty and quality improvement in critical care' consortium has already focused attention on TBI and has just started collecting additional information on this condition in order to develop a prognostic model to identify centers of excellence in TBI management. Aims of the CREACTIVE project are to consolidate the existing network in order to better describe the epidemiology of moderate-to-severe TBI in 7 countries (Cyprus, Greece, Hungary, Israel, Italy, Poland, Slovenia); establish centralized repositories of biological samples (blood and derived fluids, CSF) and clinical imaging data, to be exploit for prognostic purposes; build a prognostic model based on clinical and biological data to predict short- and long-term outcome; identify most effective clinical interventions for optimally treating TBI patients; recognize the determinants of optimal vs. suboptimal performance.

All patients admitted to the participating ICUs with a diagnosis of traumatic brain injury, regardless of their severity, will be recruited. Centralized repositories of imaging data and biological samples for the analysis of phenotypic and genotypic biomarkers will be established for approx. 2,000 adult TBI patients.

Follow-up will be performed six months after the trauma event, and will be two-tiered. The first level will be administered over the phone and constituted of the extended version of the Glasgow Outcome Scale (GOSe) and a health-related quality of care questionnaire. The second level will encompass a patient's full examination that, for children, will include a dedicated sleep disturbances study. The second level follow-up will be performed in a selected subgroup of ICUs.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the participating ICUs with a diagnosis of traumatic brain injury, regardless of their severity,will be recruited.

Exclusion Criteria:

Absence of Informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TBI patients admitted to ICU for specific care
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extendend (GOSe) | 6 months
Quality of life in Brain Injury Overall Scale (QOLIBRI-OS) | 6 months

SECONDARY OUTCOMES:
Mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (20):
- Italy (20):
  - Ospedale Regionale della Valle d'Aosta, Aosta, Aosta Valley
  - A.O. Universitaria Policlinico "Riuniti", Foggia, Apulia
  - Ospedale Santa Maria di Loreto, Napoli, Campania
  - Ospedale Maggiore, Bologna, Emilia Romagan
  - AUSL della Romagna, Ospedale Bufalini, Cesena, Emilia-Romagna
  - Ospedale San Camillo Forlanini, Rome, Lazio
  - Presidio Ospedliero di Cremon, Cremona, Lombardy
  - Niguarda Cà Granda, Milan, Lombardy
  - Ospedale A. Manzoni, Lecco, Lombradia
  - SS. Antonio e Biagio e C. Arrigo, Alessandria, Piedmont
  - Ospedale Edoardo Agnelli, Pinerolo, Piedmont
  - CTO Maria Adelaide, Turin, Piedmont
  - Ospedale Giovanni Paolo II, Olbia, Sardinia
  - AO Villa Sofia - Cervello, Palermo, Sicily
  - Ospedale San Salvatore, Pesaro, The Marches
  - Ospedale del Mugello, Borgo San Lorenzo, Tuscany
  - AO Universitaria Careggi, Florence, Tuscany
  - Ospedale di S. Chiara, Pisa, Tuscany
  - Ospedale di Santa Chiara, Pisa, Tuscany
  - Ospedale Santa Maria della Misericordia, Perugia, Umbria

REFERENCES:
- See also: Related info — http://www.giviti.marionegri.it